CLINICAL TRIAL: NCT05062252
Title: Multicentric, Prospective, Comparative Trial to Assess the Efficacy and Safety of an Anatomic Total Shoulder System.
Brief Title: Mirror Medacta Shoulder System Pivotal Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06.003.01
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Arthritis Shoulder; Post-traumatic Arthrosis of Other Joints, Upper Arm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror group (Experimental): Mirror Medacta Shoulder System
  Interventions: Device: Mirror Medacta Shoulder System
- Historical Control group (Active Comparator): Total shoulder arthroplasty system
  Interventions: Device: Medacta Shoulder System

INTERVENTIONS:
Device: Mirror Medacta Shoulder System — Anatomic total shoulder arthroplasty system
  Arms: Mirror group
Device: Medacta Shoulder System — Anatomic total shoulder arthroplasty system - standard configuration
  Arms: Historical Control group

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of the Mirror Medacta Shoulder System in total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yr
* Clinical indication for anatomic primary total shoulder replacement due to osteoarthritis and/or posttraumatic arthritis
* Willingness and ability to comply with study protocol

Exclusion Criteria:

* Medical condition or balance impairment that could lead to falls
* Prior rotator cuff surgery
* Cuff tear arthropathy/insufficient rotator cuff
* Insufficient bone quality which may affect the stability of the implant
* Neuromuscular compromise of shoulder or other disabilities affecting the maximum functional outcomes
* Weight bearing shoulder due to wheel chair, crutches, rollator at the time of operation
* Active metastatic or neoplastic disease at the shoulder joint
* Chemotherapy treatment/radiotherapy within 6 mo before surgery
* >5 mg/day of corticosteroids, excluding inhalers, within 3 years before surgery
* Pregnancy or plan to become pregnant during study period
* Inability to understand study or a history of noncompliance with medical advice
* Alcohol or drug abuse
* Current enrollment in any clinical research study that might interfere with this study
* Metal allergies or sensitivity.
* Previous or current infection at or near the site of implantation.
* Current distant or systemic infection
* Patient, whose infomed consent form should be taken in an emergency situation
* ONLY for women of childbearing age: a positive pregnancy test (urine / blood)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 12 months
  0 (worst) - 48 (best)

SECONDARY OUTCOMES:
Device Success Rate | 24 months
  Kaplan Meier survival curve, examining the following end-points:
  1. component revision for any reason;
  2. aseptic loosening;
  3. any definite change in the position of components.
Oxford Shoulder Score | 24 months
  0 (worst) - 48 (best)
Constant score | 24 months
  0(worst) - 100 (best)
Subjective Shoulder Value | 24 months
  0(worst) - 100 (best)
Device parameters | 24 months
  Devices will be assessed to determine percentage of participants that demonstrated the following after total shoulder arthroplasty:
  1. Radiolucencies,
  2. Migration,
  3. Osteolysis,
  4. Subsidence

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Zumstein, Prof Dr. med, Principal Investigator — Lindenhofgruppe AG (Bern)
Locations (2):
- Switzerland (2):
  - Lindenhofgruppe AG - Orthopädie Sonnenhof, Bern
  - Klinik für Orthopädische Chirurgie und Traumatologie des Bewegungsapparates, Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No